CLINICAL TRIAL: NCT04324554
Title: Evaluation of the Diagnostic Value of a Biomarker of Non-surgical Knee Osteoarthritis: Subchondral Bone Perfusion (GENU-PERF)
Brief Title: Diagnostic Value of a Biomarker of Non-surgical Knee Osteoarthritis
Acronym: GENU-PERF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0081
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Subchondral bone; DCE-MRI
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MRI of the right knee: An MRI of the right knee will be done to define the role of imaging in the diagnosis of early femoro-patellar osteoarthritis.
  Interventions: Diagnostic Test: MRI of the right knee

INTERVENTIONS:
Diagnostic Test: MRI of the right knee — An MRI of the right knee will be done to define the role of imaging in the diagnosis of early femoro-patellar osteoarthritis.

SUMMARY:
Osteoarthritis is a very common pathology, especially in an aging population, and a source of disability. Based on standard radiography, the diagnosis is performed late based on the loss of the cartilage thickness. In this context, prosthetic replacement of the joint is a frequent outcome. New diagnostic biomarkers and herapeutic targets are therefore logically research priorities identified by the European League Against Rheumatisms, osteoarthritis ad hoc committee. The inflammation related to the development of this pathology is mainly studied at the cellular level and essentially in animals. Since inflammatory and vascular phenomena are closely intertwined, medical imaging of the subchondral bone vascularization appears interesting.

The dynamic contrast-enhanced T1 Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) technique allows the identification of changes in the osteoarthritic subchondral bone vascularization. In osteoarthritic animals, these changes could be identified before the cartilaginous lesions became visible, and could be correlated with the severity of osteoarthritis.

This study would be the first to correlate subchondral bone perfusion measurements (performed with the DCE sequence) of early cartilaginous lesions of the knee, identified by non-invasive MRI (T2 mapping) in humans. This examination will be performed on a 3 Tesla MRI.

If a correlation is demonstrated in the early stages of osteoarthritis in both humans and animals, then infusion of subchondral bone could become a biomarker of osteoarthritis, and serve as a follow-up evaluation of future treatments.

DETAILED DESCRIPTION:
Osteoarthritis is a very common pathology, especially in an aging population, and a source of disability. Based on standard radiography, the diagnosis is performed late because it is based on the loss of cartilage thickness. In this context, prosthetic replacement of the joint is a frequent outcome. New diagnostic biomarkers and new therapeutic targets are therefore logically research priorities identified up today by the European League Against Rheumatisms, osteoarthritis ad hoc committee .

The strictly mechanical nature of osteoarthritis is currently being questioned. Indeed, the primitive role of inflammation in the development of this pathology is more and more discussed. This inflammation is today studied at the cellular level and essentially in animals. Since inflammatory and vascular phenomena are closely intertwined, medical imaging of the subchondral bone vascularization appears interesting.

The dynamic contrast-enhanced T1 Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) technique allows the identification of changes in the osteoarthritic subchondral bone vascularization. In osteoarthritic animals, these changes could be identified before the cartilaginous lesions became visible, and could be correlated with the severity of osteoarthritis.

In humans, a preliminary investigator study has recently shown that these changes correlate with the importance of osteoarthritic lesions in patients with advanced osteoarthritis. Up to date, no clinical study has so far been initiated to evaluate the diagnostic value of vascularization markers of subchondral bone in early knee osteoarthritis.

In this context, this prospective monocentric study aims to define the role of DCE medical imaging in the diagnosis of early (non-surgical) patella-femoral osteoarthritis.

This study would be the first to correlate subchondral bone perfusion measurements (performed with the DCE sequence) with early cartilaginous lesions, identified by non-invasive MRI (T2 mapping) in humans. This examination will be performed on a 3 Tesla MRI.

If a correlation is demonstrated in the early stages of osteoarthritis in both humans and animals, then infusion of subchondral bone could become a biomarker of osteoarthritis, and serve as a follow-up evaluation of future treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old and < 60 years old
* Asymptomatic at the patella-femoral joint
* Coming to perform a medical imaging examination for another indication, in the medical imaging department of the GHICL
* Patient being informed and given free, informed and written consent to participate
* Affiliated to the social security

Exclusion Criteria:

* Medical history of traumatic ligamentous, meniscal or cartilaginous lesion
* Medical history of knee surgery
* Contraindications to MRI (pacemaker, ferromagnetic vascular clip, infusion pump, neurostimulator, cochlear implant, suspicion of metallic foreign body, claustrophobia, ...)
* MRI with gadoteric acid injection in the 7 days preceding the MRI of the knee
* Hypersensitivity to gadoteric acid, meglumine or any drug containing gadolinium, or any other contrast medium
* Medical history of severe allergy, uncontrolled asthma, treatment with beta-blocker
* Renal insufficiency: glomerular filtration less than 30 mL/min
* Pregnant or nursing woman
* Patient under tutorship or curatorship

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Asymptomatic persons coming to perform a medical imaging examination for another indication, in the medical imaging department of the GHICL.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between T2 cartilage value and endothelial transfer constant (Ktrans) | Thirty minutes after MRI
  T2 (transverse relaxation time) mapping can evaluate the status of the cartilage matrix and identify biochemical changes. T2 is the time constant which determines the rate at which excited protons reach equilibrium or go out of phase with each other. It is a measure of the time taken for spinning protons to lose phase coherence among the nuclei spinning perpendicular to the main field.
  Ktrans is a constant representing the volume transfer between blood plasma and extravascular extracellular space. its units are given in values of (1/time)
Correlation between T2 cartilage value and reflux rate (Kep) | Thirty minutes after MRI
  The infusion pharmacokinetics parameters are as follows:
  Ktrans, Kep Kep represents the time constant for gadolinium reflux from the extravascular extracellular space back into the vascular system
Correlation between T2 cartilage value and initial slope of the kinetic curve | Thirty minutes after MRI
  The infusion non-pharmacokinetics parameters are as follows:
  - initial slope, time at peak, area under the curve
Correlation between T2 cartilage value and area under the kinetic curve | Thirty minutes after MRI
  The infusion non-pharmacokinetics parameters are as follows:
  - initial slope, time at peak, area under the curve
Correlation between T2 cartilage value and time at peak | Thirty minutes after MRI
  The infusion non-pharmacokinetics parameters are as follows:
  - initial slope, time at peak, area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François BUDZIK, Pr, Principal Investigator — Lille Catholic University
Locations (1):
- Lille Catholic Hospitals, Lomme, Nord, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conaghan PG, Kloppenburg M, Schett G, Bijlsma JW; EULAR osteoarthritis ad hoc committee. Osteoarthritis research priorities: a report from a EULAR ad hoc expert committee. Ann Rheum Dis. 2014 Aug;73(8):1442-5. doi: 10.1136/annrheumdis-2013-204660. Epub 2014 Mar 13. PMID 24625626
- See also: Osteoarthritis (OA) currently affects over 40 million Europeans, with its associated personal suffering and significant economic burden for health systems set to dramatically escalate in a rapidly ageing Europe. — https://ard.bmj.com/content/73/8/1442.full